CLINICAL TRIAL: NCT01783171
Title: A Phase I Trial of Dinaciclib (SCH727965) and MK-2206 in Metastatic Pancreatic Cancer With an Expansion Cohort in Advanced Pancreatic Cancer
Brief Title: Dinaciclib and Akt Inhibitor MK2206 in Treating Patients With Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00153; NCI-2013-00153 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NA_00075037; J1269; 9231 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 9231 (Other: CTEP); P30CA006973 (NIH); R21CA172997 (NIH); U01CA132123 (NIH); U01CA070095 (NIH); UM1CA186644 (NIH); UM1CA186688 (NIH); UM1CA186691 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage III Pancreatic Cancer AJCC v6 and v7; Stage IV Pancreatic Cancer AJCC v6 and v7; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — MK 2206; dinaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (dinaciclib, Akt inhibitor MK2206) (Experimental): Patients receive dinaciclib IV over 2 hours on day 1 of course 1.
  After day 1, all patients receive Akt inhibitor MK2206 PO on days 1, 8, and 15 and dinaciclib IV over 2 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Dinaciclib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm B (Akt inhibitor MK2206, dinaciclib) (Experimental): Patients receive Akt inhibitor MK2206 PO on day 1 of course 1.
  After day 1, all patients receive Akt inhibitor MK2206 PO on days 1, 8, and 15 and dinaciclib IV over 2 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Dinaciclib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
Drug: Dinaciclib — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase I trial studies the side effects and best dose of dinaciclib and Akt inhibitor MK2206 in treating patients with pancreatic cancer that cannot be removed by surgery. Dinaciclib and Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD), safety, and toxicity of the combination of MK-2206 (Akt inhibitor MK2206) and dinaciclib in patients with advanced pancreatic adenocarcinoma (Level 2.5, determined August 2015: Dinaciclib 9 mg/m2 intravenously [IV]; MK-2206 135 mg orally [PO]).

SECONDARY OBJECTIVES:

I. Assess the preliminary efficacy of the combination of MK-2206 and dinaciclib in metastatic pancreatic cancer patients as determined by disease control rate in an expansion cohort of patients at the MTD.

II. Characterize the pharmacokinetic (PK) profile of the combination of MK-2206 and dinaciclib.

III. Analyze pre-treatment tumor specimens for activation of retrovirus-associated deoxyribonucleic acid (DNA) sequence (RAS) downstream pathway signaling as potential predictors of treatment benefit.

IV. Correlate post-treatment pharmacodynamic (PD) changes in phosphorylated extracellular signal-regulated kinase (p-ERK), phosphorylated-v-akt murine thymoma viral oncogene homolog 1 (p-AKT), p-ribosomal protein S6 kinase (S6), phosphorylated DNA-directed ribonucleic acid (RNA) polymerase II subunit RPB1 (pPOLR2), phosphorylated retinoblastoma protein (pRB), proliferation-related Ki-67 antigen (Ki-67), and cleaved caspase-3 in tumor biopsies and peripheral blood mononuclear cells with MK-2206 and dinaciclib exposure and treatment response to demonstrate proof-of-concept and assess for post-treatment predictive biomarkers.

V. To assess the effect of polymorphic variations in candidate genes (cytochrome P450 3A4/5 [CYP3A4/5], ATP-binding cassette, sub-family B [MDR/TAP], member 1 [ABCB1]) and other genetic alterations that may be discovered during the conduct of the study, on MK-2206 and dinaciclib disposition, toxicity, and efficacy.

OUTLINE: This is a dose-escalation study. Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive dinaciclib IV over 2 hours on day 1 of course 1.

ARM B: Patients receive Akt inhibitor MK2206 PO on day 1 of course 1.

After day 1, all patients receive Akt inhibitor MK2206 PO on days 1, 8, and 15 and dinaciclib IV over 2 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed, unresectable pancreatic adenocarcinoma
* Patients must have already received or refused 1st-line treatment
* Measurable disease will be required; biopsiable disease will be required
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 16 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X IULN if no liver metastasis or =< 5 X IULN if liver metastases are present
* Creatinine not to be above IULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MK-2206 and dinaciclib administration
* Patients must be able to swallow whole tablets (for MK-2206); nasogastric or gastrostomy (G) tube administration is not allowed; tablets must not be crushed or chewed
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to =< grade 1 (or =< tolerable grade 2 for neuropathy) adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dinaciclib or to MK-2206
* Patients receiving any medications or substances that are strong inhibitors/inducers, sensitive substrates, or substrates with a narrow therapeutic index of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) or permeability glycoprotein (P-gp) are ineligible; caution should be exercised when dosing dinaciclib and/or MK-2206 concurrently with CYP3A4 or P-gp substrates, inhibitors/inducers; if subjects are taken off a forbidden medicine, a one-week washout is required for inhibitors and two weeks for inducers; subjects on Coumadin are eligible but more frequent monitoring of the international normalized ratio (INR) (weekly during the first cycle, then at least each cycle thereafter) is recommended; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled before the patient enters the trial (glycosylated hemoglobin [Hba1c] < 7.5)
* Concurrent medications associated with a risk of corrected QT (QTc) prolongation and/or torsades de pointes are not allowed; those medications listed as reported but lacking substantial evidence for causing QTc prolongation and torsades de pointes will be allowed, although if an alternative medication can be substituted, that would be preferable; for this study, a baseline electrocardiogram (EKG) will be performed and will be repeated during cycle 1 and then every 3 cycles while on treatment
* Patients with current evidence of significant cardiovascular disease (New York Heart Association class III or IV cardiac disease), symptomatic congestive heart failure, dilated/hypertrophic or restrictive cardiomyopathy, myocardial infarction (within the past 6 months), unstable angina, unstable arrhythmia or a need for anti-arrhythmic therapy (use of medications for rate control for atrial fibrillation is allowed such as calcium channel blockers and beta-blockers, if stable medication for at least last month prior to initiation of MK-2206 treatment and medication not listed as causing torsades de pointes), or evidence of acute ischemia on electrocardiogram (ECG); marked baseline prolongation of QT/QTc interval, e.g., repeated demonstration of a QTc interval > 450 msec*; long QT syndrome; the required use of concomitant medication that may cause torsades de pointes or may cause a significant prolongation of the QTc

  * Note: Due to difficulties assessing QTc in patients with heart block, they may be eligible if deemed safe by a cardiologist
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK-2206 and/or dinaciclib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Clinically significant ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
MTD of dinaciclib in combination with Akt inhibitor MK2206 defined as the highest dose at which 0 or 1 dose-limiting toxicities are observed in six patients | 28 days
  The proportion of dose-limiting toxicities at each dose level will be reported with exact binomial proportions and 95% confidence intervals.

SECONDARY OUTCOMES:
Disease control rate: complete response, partial response and stable disease evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1 | 4 months
  Calculated with exact 95% confidence intervals. The exact Cochran-Armitage trend test will be used to test if the probability of controlled disease at four months is increased with combinations of greater baseline activation of Ras and greater inhibition of Ras downstream pathway signaling. Logistic regression will be used to assess the effects of multiple covariates on the probability of controlled disease at 4 months.
Incidence of adverse events of the combination of dinaciclib and Akt inhibitor MK-2206, graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 1 year
  The proportion of toxicities by type and grade will be reported with exact binomial proportions and 95% confidence intervals. Adverse events will be summarized by dose level for all doses.
Overall survival | Up to 1 year
  Summarized using overall hazard rate estimates and 95% confidence intervals as well as Kaplan-Meier (KM) estimates.
Progression-free survival | Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
  Summarized using overall hazard rate estimates and 95% confidence intervals as well as KM estimates. The median PFS and median survival will be reported. Cox proportional hazards models will be used to evaluate the impact of key covariates on PFS and survival.

OTHER OUTCOMES:
Change in protein expression in serum after treatment with a single drug, and after treatment with both drugs as a measure of the drug specific effects on pathway markers | Baseline up to day 3 of course 2
Change in protein expression in the tumor tissue before and after treatment using semi-quantitative immunohistochemical (IHC) analysis as a measure of response to therapy | Baseline up to day 3 of course 2
Inhibition and concordance of cyclin-dependent kinase (CDK)/Ral and phosphatidylinositol 3 kinase (PI3K)/pAkt pathways as measured in serum and tissue samples | Up to day 3 of course 2
  Inhibition of the CDK/Ral pathway with dinaciclib will be assessed by pRb and pPOLR2, while inhibition of the downstream PI3K/pAkt pathway with MK-2206 will be evaluated with pAkt and pS6. A summary score will be obtained for each pathway by summing the HistoScores of the markers in that pathway. The percent inhibition of each pathway will be calculated as the percentage decrease in the summary score, relative to the pre treatment score. The concordance of the inhibition of both pathways, as measured in the serum samples, and as measured in the tissue, will be assessed with Kappa statistic.
Pharmacokinetic profile of the combination of Akt inhibitor MK-2206 and dinaciclib | Pre-dose, at start of dinaciclib infusion, 5 minutes prior to end of dinaciclib infusion, 0.5, 1, 1.5, 2, 4, and 8 hours after end of dinaciclib infusion on day 1 of course 1; at 24, 48, and 96 hours after Akt inhibitor MK-2206 infusion; days 8 and 15
  Will summarize and analyze the data via two-by-two tables, separately for each drug. Total exposure on each day will be calculated as area under the plasma concentration-time curve (AUC) using the linear or log-linear trapezoidal rule by using noncompartmental methods and/or compartmental modeling. Maximum concentration (Cmax) and time to maximal concentration (Tmax) and minimum or trough concentrations (Cmin) will be obtained from the observed data.
Polymorphic variations in candidate genes (CYP3A4/5, ABCB1) | Up to day 3 of course 2
  Other genetic alterations that may be discovered during the conduct of the study, on MK-2206 and dinaciclib disposition, toxicity, and efficacy will be assessed.
Protein expression in serum as measured by fluorescence activated cell sorting (FACS) | Up to day 3 of course 2
  The correlation of serum pathway markers and these same markers measured in tissue samples with IHC will be assessed using Spearman's correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (5):
- United States (4):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hu C, Dadon T, Chenna V, Yabuuchi S, Bannerji R, Booher R, Strack P, Azad N, Nelkin BD, Maitra A. Combined Inhibition of Cyclin-Dependent Kinases (Dinaciclib) and AKT (MK-2206) Blocks Pancreatic Tumor Growth and Metastases in Patient-Derived Xenograft Models. Mol Cancer Ther. 2015 Jul;14(7):1532-9. doi: 10.1158/1535-7163.MCT-15-0028. Epub 2015 Apr 30. PMID 25931518